CLINICAL TRIAL: NCT06843772
Title: Investigation of the Relationship Between Digital Game Addiction and Musculoskeletal System Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar22
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Game Addiction, Video
MeSH Terms: conditions — Technology Addiction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): People who do not have any exercise program
  Interventions: Other: ergonomic training
- exercise (Experimental): People who will have an exercise program
  Interventions: Other: ergonomic training; Other: exercise

INTERVENTIONS:
Other: ergonomic training — will receive ergonomic training.
Other: exercise — People who will receive an exercise program. Participants will receive ergonomic training along with the exercise program.
  Arms: exercise

SUMMARY:
The aim of this study is to examine the effects of digital game addiction on the musculoskeletal system and the reflections of these effects on the quality of life of adults.

DETAILED DESCRIPTION:
This study will be conducted with a cross-sectional design in order to examine the relationship between digital game addiction and musculoskeletal disorders. The methods to be used in the research are as follows: Participant Information: The study will include adults aged 18-39 who play digital games in internet cafes for at least 3 hours a day, 4-5 days a week. Participants will be asked to fill out a form to collect demographic information. This form will include information such as age, gender, weekly game playing frequency (by hour and day), and physical activity levels. Scales to be Used: The following measurement tools will be used in the study to evaluate the effects of digital game addiction on the musculoskeletal system. Digital Game Addiction Scale, Arm, Shoulder and Hand Problems Questionnaire, Pittsburgh Sleep Quality, Cornell Musculoskeletal Disorder Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-39.
* Individuals who play digital games at least 4-5 days a week, at least 3 hours a day.
* Individuals who voluntarily participate in the study and sign the ethical consent form.

Exclusion Criteria:

* Individuals with existing serious health problems related to the musculoskeletal system or sleep patterns.
* Individuals who suffered trauma or serious injuries related to the musculoskeletal system during the study period.
* Individuals with psychological disorders such as depression or anxiety disorder.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Disorder Questionnaire | 14 weeks
  The questionnaire was conducted in 11 body regions (neck, right and left shoulder, upper arm, forearm and wrist, back and waist region) includes questions about the frequency of musculoskeletal disorders (pain/pain/discomfort), the severity of these disorders, and whether they interfere with work.
The Pittsburgh Sleep Quality Index | 14 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".
Disabilities of the Arm, Shoulder and Hand Questionnaire | 14 weeks
  It was developed to evaluate functional status and symptoms by focusing on physical function in upper extremity injuries. According to the results of the survey; a result from 0-100 is obtained from each part; 0-no apology 100-maximum apology.

CONTACTS AND LOCATIONS:
Overall Officials: Lobaba Chiah, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed S, Samuel AJ, Mishra A, Rahman MS, Islam MA, Rashaduzzaman M, Roy SK, Akter R, Islam MJ. Mobile game addiction and its association with musculoskeletal pain among students: A cross-sectional study. PLoS One. 2024 Aug 26;19(8):e0308674. doi: 10.1371/journal.pone.0308674. eCollection 2024. PMID 39186761
- [Background] Brevers D, King DL, Billieux J. Delineating adaptive esports involvement from maladaptive gaming: a self-regulation perspective. Curr Opin Psychol. 2020 Dec;36:141-146. doi: 10.1016/j.copsyc.2020.07.025. Epub 2020 Aug 3. PMID 32795945
- [Background] Gulu M, Yagin FH, Gocer I, Yapici H, Ayyildiz E, Clemente FM, Ardigo LP, Zadeh AK, Prieto-Gonzalez P, Nobari H. Exploring obesity, physical activity, and digital game addiction levels among adolescents: A study on machine learning-based prediction of digital game addiction. Front Psychol. 2023 Mar 3;14:1097145. doi: 10.3389/fpsyg.2023.1097145. eCollection 2023. PMID 36936011